CLINICAL TRIAL: NCT06468150
Title: Mechanical Thrombectomy and Catheter Directed Thrombolysis Utilization in Patients With Deep Vein Thrombosis
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Igor Zolotukhin, Professor of Surgery, Pirogov RNRMU, Zolotukhin Igor Anatolievich, Pirogov Russian National Research Medical University
Other Study IDs: 224/22
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Deep Vein Thrombosis
Keywords: Mechanical thrombectomy; catheter directed thrombolysis; iliofemoral deep vein thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the utilization of mechanical thrombectomy and catheter-directed thrombolysis in patients with deep vein thrombosis in tertiary care. The main questions it aims to answer are:

1. How many patients with deep vein thrombosis are potentially eligible for mechanical thrombectomy and catheter-directed thrombolysis in a tertiary hospital?
2. What is the actual number of patients undergoing endovascular interventions for deep vein thrombosis?

Participants received endovascular treatment according to the clinical protocol of the treatment.

DETAILED DESCRIPTION:
Tertiary hospital database was analyzed. All the records of patients referred for deep vein thrombosis were extracted. The collected data included general patient information, medical history, results of physical examination, duplex ultrasound, laboratory analysis, etc. Indications and contraindications for mechanical thrombectomy and catheter-directed thrombolysis were assessed, considering possible benefits and risks. Patients who could be eligible for this technique were identified

ELIGIBILITY:
Inclusion Criteria:

* lower limb, pelvic, or inferior vena cava deep vein thrombosis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with deep vein thrombosis referred to the hospital from January 2022 to December 2023.
Sampling Method: Probability Sample
Enrollment: 2427 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with deep vein thrombosis who could be eligible for mechanical thrombectomy and catheter-directed thrombolysis | from date of admission until the date of discharge, up to 1-2 weeks
  The number of participants with deep vein thrombosis who would fit the eligibility criteria for performing the intervention

SECONDARY OUTCOMES:
The number of patients with deep vein thrombosis who underwent mechanical thrombectomy and catheter-directed thrombolysis | from date of admission until the date of discharge, up to 1-2 weeks
  The number of participants with deep vein thrombosis who fitted the eligibility criteria and underwent the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation, Moscow, Russia